CLINICAL TRIAL: NCT02709187
Title: DP-R208 Pharmacokinetic Study Phase I
Brief Title: DP-R208 Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DP-CTR208-I-04
Record Dates: First submitted 2016-02-17; First posted 2016-03-15 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: DP-R208
MeSH Terms: interventions — candesartan cilexetil; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RT group (Experimental): combination dose of Candesartan and Rosuvastatin and DP-R208 in order
  Interventions: Drug: DP-R208; Drug: Candesartan cilexetil; Drug: Rosuvastatin
- TR group (Experimental): DP-R208 and combination dose of Candesartan and Rosuvastatin in order
  Interventions: Drug: DP-R208; Drug: Candesartan cilexetil; Drug: Rosuvastatin

INTERVENTIONS:
Drug: DP-R208 — Investigational product is prescribed to all of randomized subjects
Drug: Candesartan cilexetil — Investigational product is prescribed to all of randomized subjects
Drug: Rosuvastatin — Investigational product is prescribed to all of randomized subjects

SUMMARY:
An open label, randomized, 2-sequence, 2-period, single-dose cross-over study to evaluate the pharmacokinetics characteristics of DP-R208 (Candesartan cilexetil 8mg/Rosuvastatin 10mg), a fixed dose combination compared with coadministration of separate constituents in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* BMI 18~30
* signed the informed consent form prior to the study participation

Exclusion Criteria:

* Clinically significant disease
* Previously donate whole blood within 60 days or component blood within 14 days
* Clinically significant allergic disease
* Taken IP in other trial within 90 days
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | up to 48 hours post dose
Peak Plasma Concentration (Cmax) | up to 48 hours post dose